CLINICAL TRIAL: NCT02653781
Title: Implementation of Realistic Simulation as Patient Safety Improvement Method: Controlled Trial
Brief Title: Implementation of Realistic Simulation as Patient Safety Improvement Method
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Marcia Cristina da Silva Magro, PhD, University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ECR222015
Record Dates: First submitted 2015-12-17; First posted 2016-01-12 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Compliance Behavior
MeSH Terms: conditions — Patient Compliance | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Realistic simulation; Performance (Experimental): Student participation in the study will happen on demand by enrollment in activities of dialogue-exhibition (workshop) on realistic simulation in the context of patient safety. Check the performance of students in face of simulation workshop for test realistic simulation.
  Interventions: Behavioral: Realistic simulation; Behavioral: control group; Behavioral: Simulation workshop; Behavioral: Test realistic simulation
- theoretical-practical classes (Other): Will be to give a theoretical-practical classes for students of control group the provision of similar opportunities
  Interventions: Behavioral: control group; Behavioral: Test realistic simulation

INTERVENTIONS:
Behavioral: Realistic simulation — The students enrolled and selected according to the inclusion criteria will be randomized into two groups. The experimental group will experience the combined teaching methodology: dialogue-exhibition and realistic simulation.
  Arms: Realistic simulation; Performance
Behavioral: control group — The control group will have contents exposed solely from the dialogue-exhibition.
Behavioral: Simulation workshop — Check the performance of students in face of simulated situations on medication administration by intramuscular and intravenous routes experienced in the Skills and Care Simulation Laboratory.
  Arms: Realistic simulation; Performance
Behavioral: Test realistic simulation — Occurs after the end of the three-month intervention. At that time, students from the control and intervention groups will be asked to take a knowledge retention test in cognitive assessment format and OSCE format (objective structured clinical examination).

SUMMARY:
Realistic simulation is an effective teaching strategy for the acquisition and retention of knowledge and increased self-confidence of students, which contribute to safety in performing nursing actions.Considering the need to adopt safe practices in health since professional training, there are deficiencies in health teaching and weaknesses in the acquisition of practical skills guided by safety principles and critical clinical reasoning. The purpose is to compare the use of high fidelity simulation with traditional education as innovative method in the process of teaching and learning. This is a prospective, randomized, controlled and single-blind study, of pre-test and post-test experimental type, with application of high fidelity simulation in the theme of patient safety in administration of parenteral drugs.

DETAILED DESCRIPTION:
Currently, the issue of patient safety has been hotly debated both nationally and internationally, because this is a relevant issue for the health professionals' practice and to improve the quality of patient care. According to the Institute of Medicine (IOM) report released in 2000, a significant number of deaths in hospitals every year were related to preventable causes and medical errors. These deaths were equal to mortality numbers due to diseases such as cancer and HIV and car acidentes.

In this scenario, death due to errors in the process of care achieved world relevance and in 2002, the World Health Organization (WHO) released the World Health Assembly (WHA) Resolution 55.18, addressing the priorities related to patient safety in the quality of care. In 2004, was created the World Alliance for Patient Safety on the occasion of the 57th World Health Assembly. The World Alliance has defined programs for patient safety that must be adopted by all member countries and therefore, by Brazil.

The general actions proposed by the WHO World Alliance for Patient Safety are oriented in five activities among which, the efforts to strengthen the training in patient safety worldwide. It stimulates the inclusion of a curriculum guide for patient safety in health professional training courses .

Aspects of patient safety in medicine administration involve many health professionals. However, nurses have an important role because they are responsible for administration and thus, occupy the last stage between the medication and the error. For all these reasons, safety in medication administration is a compulsory and transversal theme in the training of nursing professionals.

In this context of search for improvements in health care planning, a new practice concept of teaching and learning has been developed, aiming at training professionals and training the health professionals who have already graduated.

Interests in using realistic simulation techniques have emerged lately with the objective to encourage improvements in safety on patient care. The simulation technique amplifies the experience of health professionals through educational actions guided by experiences that happen in the real world, therefore, interactions must happen in a way that preserves the most realistic aspects as possible. The adoption of simulation in health comes from successful references of using this technique for industrial purposes and in the armed forces. It is considered an innovative technique in health.

In high fidelity simulation, students and professionals experience clinical cases that replicate real-world scenarios. This strategy enables teaching innovations, improves clinical thinking in stressful situations, and prevents the exposure of patients to risks.

The realistic simulation has been integrated in the education of nurses and doctors over the last years, but is not fully implemented yet. Despite the recommendations for using simulation, its increasing integration in education, and the concrete evidence that its use promotes a better prepare of health professionals for performance in clinical practice, the empirical evidences of its impact on patient outcomes are still under developed.

Besides the realistic manikin-based simulation, virtual simulation is another way of simulation that has been proven effective in learning strategies, contributing to the retention of knowledge and improvement of nursing students' clinical performance.

From the increasing use of technology in health and the complexity of patients, new ways of learning have been shaped and developed as innovative teaching methods in health care . All these alternatives have the promising intention of reducing the deterioration of learning and of clinical performance over time, making professionals and students able to monitor patients in the best possible way, establish goals, priorities and better treatments.

An advantage is the possibility of students practicing their skills in an environment where mistakes can be made and corrected without causing damages and risks to patient safety. In addition, the construction of knowledge is established through representative situations of day-to-day reality in professional practice, when students themselves participate as patient-actors in a totally controlled environment, as well as protected from risks. At the end of the activity, students and/or professionals involved in the simulation can give feedback of their learning and, from group discussions and those with the teacher, is formed knowledge based on self-knowledge and confidence .

PURPOSE

Primary purpose

To compare the use of high fidelity simulation with traditional education as innovative method in the process of teaching and learning.

Secondary purpose

To propose the creation of a high fidelity scenario related to nursing care in medication administration;

To identify the gains in theoretical and practical learning and in self-confidence of nursing undergraduate students after undergoing high fidelity simulation in medication administration;

To assess the effectiveness and efficiency of using high fidelity simulation in the process of teaching and learning.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Regularly enrolled in the nursing undergraduate course at the Universidade de Brasília - Ceilândia Institute
* Attending between the sixth and tenth semester of the nursing undergraduate course at the Universidade of Brasília
* Already took the 'Semiology I' discipline

Exclusion Criteria:

* Less than 18 years
* Student with another formation of secondary or higher level in the area of victims service or health care (eg: nursing technician, firefighter, paramedic, physical therapist, etc)
* Missing at least one of the study steps: pre-test, workshop, post-test, experience in realistic simulation, retest

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness assessed using questionnaire and scale with the scores range from 0 (no effectiveness) to 5 (with effectiveness) | The outcome measures are assessed as up to six months rather than the specific dates provided
  Assess the effectiveness of using high fidelity simulation in the process of teaching and learning using questionnaire and scale with the scores range from 0 (no effectiveness) to 5 (with effectiveness)

SECONDARY OUTCOMES:
Efficiency assessed by using questionnaire and scale from 0 (no efficiency) to 5 (with efficiency) | The outcome measures are assessed as up to six months rather than the specific dates provided
  Assess the efficiency of using high fidelity simulation in the process of teaching and learning until for 3 months later to begin the study with questionnaire and scale from 0 (no efficiency) to 5 (with efficiency)

OTHER OUTCOMES:
Gains in theoretical learning and in self-confidence of nursing assessed using a scale from 0 to 5. | The outcome measures are assessed as up to six months rather than the specific dates provided
  To identify the gains in theoretical learning and in self-confidence of nursing undergraduate students after undergoing high fidelity simulation in medication administration using scale from 0 to 5.
Gains in practical learning and in self-confidence of nursing assessed using a scale from 0 to 5. | The outcome measures are assessed as up to six months rather than the specific dates provided
  To identify the gains in practical learning and in self-confidence of nursing undergraduate students after undergoing high fidelity simulation in medication administration using scale from 0 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Cristina S. Magro, PhD, Principal Investigator — Brasilia University

REFERENCES:
- [Background] Aebersold M, Tschannen D. Simulation in nursing practice: the impact on patient care. Online J Issues Nurs. 2013 May 31;18(2):6. PMID 23758424
- [Background] Boutron I, Moher D, Altman DG, Schulz KF, Ravaud P; CONSORT Group. Extending the CONSORT statement to randomized trials of nonpharmacologic treatment: explanation and elaboration. Ann Intern Med. 2008 Feb 19;148(4):295-309. doi: 10.7326/0003-4819-148-4-200802190-00008. PMID 18283207
- [Background] Frith KH, Anderson EF, Tseng F, Fong EA. Nurse staffing is an important strategy to prevent medication error in community hospitals. Nurs Econ. 2012 Sep-Oct;30(5):288-94. PMID 23198612
- [Background] Gaba DM. The future vision of simulation in health care. Qual Saf Health Care. 2004 Oct;13 Suppl 1(Suppl 1):i2-10. doi: 10.1136/qhc.13.suppl_1.i2. PMID 15465951
- [Background] Godson NR, Wilson A, Goodman M. Evaluating student nurse learning in the clinical skills laboratory. Br J Nurs. 2007 Aug 9-Sep 12;16(15):942-5. doi: 10.12968/bjon.2007.16.15.24520. PMID 17851322
- [Background] Harden RM, Gleeson FA. Assessment of clinical competence using an objective structured clinical examination (OSCE). Med Educ. 1979 Jan;13(1):41-54. No abstract available. PMID 763183
- [Background] Jeffries PR, McNelis AM, Wheeler CA. Simulation as a vehicle for enhancing collaborative practice models. Crit Care Nurs Clin North Am. 2008 Dec;20(4):471-80. doi: 10.1016/j.ccell.2008.08.005. PMID 19007713
- [Background] Lewis R, Strachan A, Smith MM. Is high fidelity simulation the most effective method for the development of non-technical skills in nursing? A review of the current evidence. Open Nurs J. 2012;6:82-9. doi: 10.2174/1874434601206010082. Epub 2012 Jul 27. PMID 22893783
- [Background] Liaw SY, Chan SW, Chen FG, Hooi SC, Siau C. Comparison of virtual patient simulation with mannequin-based simulation for improving clinical performances in assessing and managing clinical deterioration: randomized controlled trial. J Med Internet Res. 2014 Sep 17;16(9):e214. doi: 10.2196/jmir.3322. PMID 25230684